CLINICAL TRIAL: NCT04292678
Title: The Effect of Progressive Relaxation Exercise on Caregiver Burden, Fatigue and Quality of Life in Caregivers of Patients With Advanced Cancer: Randomized Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Gulbahar, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N/Y
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Caregiver Burnout; Cancer
Keywords: Caregiver burden, fatigue, relaxation, quality of life.
MeSH Terms: conditions — Caregiver Burden; Neoplasms; Fatigue | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation (Experimental): Caregivers of patients with advanced cancer will apply 20 minutes of progressive muscle relaxation exercise twice a week, for 8 weeks with a group session.
  Interventions: Behavioral: Progressive muscle relaxation
- Attention matched control (Active Comparator): Caregivers of patients with advanced cancer will receive only a training group session about general cancer information such as risk factors, treatment methods, and treatment-related side effects, lasting 20 minutes first week of the study.
  Interventions: Other: Attention matched control

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — The progressive muscle relaxation intervention will last for 20 minutes and comprise sessions involving tensing and relaxing the body with deep breathing. The participants will perform progressive muscle relaxation for each body part in order, starting with the facial muscles and head, followed by neck, shoulders, chest, abdomen, legs, and feet; all muscle tension and relaxation procedures were performed accompanied with deep breathing. The participants will be instructed to tense a specified group of muscles for 5 s and relax it for 10 s while breathing out. Throughout this exercise, the participants will visualize a wave of relaxation flowing over their body using the deep-breathing technique.
  Arms: Relaxation
Other: Attention matched control — Caregivers of patients with advanced cancer will receive only a training group session about general cancer information such as risk factors, treatment methods, and treatment-related side effects, lasting 20 minutes first week of the study.
  Arms: Attention matched control

SUMMARY:
Caregivers of patients with advanced cancer will be entered. Participants will be randomized to one of two study arms: Arm 1: Progressive muscle relaxation; Arm 2: Attention matched control. Hypothesis: Progressive muscle relaxation will decrease caregiving burden and severity of fatigue and improve quality of life.

DETAILED DESCRIPTION:
Previous reports have revealed that progressive muscle relaxation to use to decrease symptom burden associated with cancer. However, there have been limited studies that directly focus on supporting caregivers of advanced cancer patients who face serious problems in diagnosis and treatment process, at least as much as cancer patients. Besides, till date, no study has been conducted to determine the effects of progressive relaxation exercise on caregiver burden, fatigue and quality of life in those providing care for patients with advanced cancer. The present study investigates the effects of progressive muscle relaxation in a single-site, 2-arm, randomized, controlled study of 64 caregivers of patients with advanced cancer. Arm 1: relaxation; Arm 2: Attention matched control. The investigators hypothesize that progressive muscle relaxation will decrease severity of caregiver burden and fatigue and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Providing care for advanced cancer patients (stage III-IV) for at least 6 months
* Primary caregiver (caring for the longest time)
* No communication problem
* Not using any other non-pharmacological approach during the study period

Exclusion Criteria:

* Providing care for individuals with early-stage (Stage I-II) cancer
* Caregivers who providing care services for a fee
* Having a history of psychiatric disorder (major depression, etc.)
* Not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver burden severity | Baseline measurements, at the end of 8th week and two weeks after the completion of the interventions
  Caregiver burden severity will be measured based on patient report by Experience-Based Caregiver Burden Scale in Advanced Cancer.
  Maximum scores indicate worse caregiver burden.
Change in fatigue severity | Baseline measurements, at the end of 8th week and two weeks after the completion of the interventions
  Fatigue severity will be measured based on patient report by the Fatigue Severity Scale. Minimum scores indicate better level of fatigue.
Change in Quality of life status | Baseline measurements, at the end of 8th week and two weeks after the completion of the interventions
  Quality of life will be measured by the Caregiver's Quality of Life Index-Cancer Scale. Maximum scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Gok Metın, Assos.Prof., Study Director — Hacettepe University

IPD SHARING:
Plan to Share IPD: No